CLINICAL TRIAL: NCT00872131
Title: Neuro-Genetic Markers of SSRI Treatment Response in Social Anxiety Disorder
Brief Title: Identifying Brain and Genetic Markers of Sertraline Treatment Response in People With Social Anxiety Disorder
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, K. Luan Phan, Associate Professor, University of Michigan
Other Study IDs: K23MH076198 (NIH); K23MH076198 (NIH); DAHBR 9A-ASPI; 5K23MH076198 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Social Phobia; Generalized Social Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Generalized social anxiety disorder participants: Participants with generalized social anxiety disorder will undergo MRI scanning and sertraline treatment.
  Interventions: Drug: Sertraline
- Healthy control participants: Healthy control participants will undergo MRI scanning.

INTERVENTIONS:
Drug: Sertraline — Oral sertraline will begin at 50 mg per day, then increase to 75 mg per day on Day 8, then increase to 100 mg per day on Day 15. The dose may be increased to 150 mg per day on Week 8, based on clinical response and medication toleration.
  Other Names: Zoloft
  Groups: Generalized social anxiety disorder participants

SUMMARY:
This study will attempt to identify gene and brain activity markers that predict whether people with social anxiety disorder will respond to selective serotonin reuptake inhibitor medications.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is an anxiety disorder characterized by excessive fear and avoidance of social situations. Selective serotonin reuptake inhibitors (SSRIs) are a medication commonly prescribed to treat social anxiety disorder, but as many as 50% of people with SAD do not respond to SSRIs. Current theory suggests that neurological functioning and genetics may influence a patient's response to treatment. This study will examine variations in genetics and brain reactivity among people with SAD who do and do not respond to SSRIs. Through this, the study will identify neurological and genetic biomarkers that can predict responsiveness to SSRI treatment in people with SAD.

Participation in this study will last 14 weeks. Both healthy people and people with SAD will be recruited to participate. All participants will complete similar study visits at entry, within 2 weeks of entry, and 12 weeks after that. The first visit, which will occur at study entry, will include screening questionnaires, an interview with research staff, a medical screening, a urine test, and collection of saliva samples for genotyping. The second visit and the last visit, which will be separated by 12 weeks, will involve MRI scans and behavioral tasks to be conducted inside and outside the MRI scanner. Over the 12 weeks between MRI scanning sessions, participants with SAD will take sertraline, a common SSRI, on a daily basis. They will also attend five additional visits during this time to complete assessments of their symptoms. These visits will occur 1, 2, 4, 8, and 12 weeks after starting sertraline treatment. Participants with SAD will therefore be completing a symptom assessment, MRI scans, and behavioral tasks all on the final visit, 12 weeks after the second visit.

ELIGIBILITY:
Inclusion Criteria:

For social anxiety disorder group:

* Current diagnosis of social anxiety disorder, generalized subtype
* Physically healthy, as confirmed by comprehensive medical history, physical exam, and laboratory testing

For healthy control group:

* Never been diagnosed with either Axis I or Axis II mental disorders
* Physically healthy, as confirmed by comprehensive medical history, physical exam, and laboratory testing

Exclusion Criteria:

* Clinically significant medical or neurologic condition
* Diagnosis of primary comorbid anxiety disorder, defined by which disorder is the more debilitating and clinically salient
* History of bipolar disorder or schizophrenia
* Presence of an organic mental syndrome, mental retardation, or pervasive developmental disorder
* Current major depressive disorder or major depression within the past 6 months
* Hamilton Rating Scale for Depression score greater than 18
* Alcohol or drug abuse or dependence within the past year
* Current suicidal ideation
* Diagnosis of an Axis II personality disorder, except for avoidant personality disorder
* Treatments with psychotropic or psychoactive medications within the 2 weeks before screening (or 8 weeks for fluoxetine and 4 weeks for monoamine oxidase inhibitors)
* Positive urine drug screen results
* Pregnancy

Additional exclusion criteria for the functional MRI studies:

* Left-handedness, as determined by standard questionnaire
* Presence of ferrous-containing metals within the body, such as aneurysm clips, shrapnel, or retained particles
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community and outpatient clinic samples
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) Scale | Measured before treatment, at five treatment study visits, and 12 weeks after starting treatment

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Measured before treatment, at five treatment study visits, and 12 weeks after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: K. Luan Phan, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States